CLINICAL TRIAL: NCT05198557
Title: Phase 3 Study of MT-0551 in Patients With Systemic Sclerosis (Placebo-Controlled Double-Blind Study)
Brief Title: A Study of MT-0551 in Patients With Systemic Sclerosis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-0551-A-301
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — inebilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MT-0551 group (Experimental): Participants will receive intravenous (IV) inebilizumab on Day 1 and Day 15 of randomized controlled period (RCP). The participants who entered open label period (OLP) will receive IV inebilizumab on Day 1 and IV placebo on Day 15 of OLP and will be followed by IV inebilizumab every 26 weeks.
  Interventions: Drug: Inebilizumab; Drug: Placebo
- Placebo group (Placebo Comparator): Participants will receive IV placebo on Day 1 and Day 15 of the RCP. The participants who entered OLP will receive IV inebilizumab on both Day 1 and Day 15 in OLP and will be followed by IV inebilizumab every 26 weeks.
  Interventions: Drug: Inebilizumab; Drug: Placebo

INTERVENTIONS:
Drug: Inebilizumab — Participants will receive IV inebilizumab.
  Other Names: MT-0551
Drug: Placebo — Participants will receive IV placebo matched to inebilizumab.

SUMMARY:
The study will verify the superiority of MT-0551 to placebo at 26 weeks after treatment initiation in systemic sclerosis (SSc) patients using the modified Rodnan Total Skin thickness Score (mRTSS) as a measure of skin thickening. The safety and pharmacokinetics will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

Additional screening criteria check may apply for qualification:

1. ACR/European League Against Rheumatism (EULAR) criteria (2013) systemic sclerosis (SSc) diagnostic criteria satisfied.
2. Skin thickening score based on the mRTSS between 10 and 22 inclusive.

Exclusion Criteria:

Additional screening criteria check may apply for qualification:

1. Pulmonary hypertension associated with SSc.
2. Presence of a serious, SSc-related concurrent illness other than interstitial pneumonia.
3. Finding of inadequate respiratory reserve capacity.
4. Past history of rituximab, blinatumomab, obinutuzumab, or ofatumumab.
5. Presence of a clinically significant active infection requiring antimicrobial therapy.
6. A past history of cancer.
7. Past history of a recurrent, clinically significant infection.
8. Past history of severe allergy or anaphylactic reaction to a biologic drug product.
9. Treatment with live vaccine within a certain period (inactivated vaccine is acceptable).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the mRTSS up to the end of the long-term extension period | baseline, RCP 4, 12, 26, OLP 4,12, 26, the long-term extension period 26, 52, 78, 104 weeks

SECONDARY OUTCOMES:
Pulmonary function tests: Change from baseline in the percent predicted forced vital capacity (%FVC) and percent predicted diffusing capacity of the lung carbon monoxide (%DLco) | Baseline to at least 52 weeks or early termination
Pulmonary function tests: Percentage change from baseline in the %FVC and %DLco | Baseline to at least 52 weeks or early termination
Change from baseline in the mRTSS | Baseline to at least 52 weeks or early termination
Composite response index in diffuse cutaneous systemic sclerosis | Week 26 to at least 52 weeks or early termination

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (4):
- Japan (4):
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - St. Marianna University Hospital, Kawasaki-shi, Kanagawa
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No